CLINICAL TRIAL: NCT06927596
Title: A Retrospective Study on the Efficacy of Interventional Treatment for Bronchopleural Fistula Related to Pulmonary Metastasis of Osteosarcoma
Brief Title: A Look Back at How Well Interventional Treatments Work for Bronchopleural Fistulas in Patients With Lung Metastases From Osteosarcoma
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-173
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Osteosarcoma Metastatic
Keywords: Pulmonary metastasis of osteosarcoma; Interventional therapy; Bronchopleural fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional THERAPY Group: Patients undergoing interventional therapy
  Interventions: Procedure: Interventional therapy

INTERVENTIONS:
Procedure: Interventional therapy — The fistula was occluded by coil and NBCA glue.

SUMMARY:
Patients with pulmonary metastasis of osteosarcoma complicated with BPF often suffer from massive hemoptysis, refractory pneumothorax and difficult fistula healing due to tumor erosion of bronchial arteries. Traditional interventional embolization (such as simple coil or gelatin sponge embolization) has some limitations such as embolic material displacement, incomplete fistula closure and postoperative recurrent bleeding. Systemic chemotherapy and radiotherapy also have poor efficacy due to the complex blood supply of local lesions and poor tissue repair ability, and the quality of life of patients is seriously impaired. Therefore, there is an urgent need to explore a safer and durable precise embolization scheme.

NBCA combined with coil closure is expected to break through the current technical bottleneck through the synergistic mechanism of "colloid embolization + mechanical occlusion". NBCA glue can quickly polymerize to achieve permanent occlusion of the micro vascular network, while the coil can strengthen the fistula through physical support. The combination of the two can not only accurately block abnormal blood supply, promote fistula healing, but also reduce the risk of embolus displacement and hemoptysis recurrence rate. This study is the first to systematically evaluate the efficacy and safety of this combination regimen in such patients, and provide key evidence for optimizing the embolization strategy and improving the long-term prognosis.

The clinical transformation value and social significance of this study are significant. If NBCA combined with coil is proved to be effective in controlling bleeding, shortening fistula closure time and reducing complications, it will promote this technology to become the first choice for advanced osteosarcoma pulmonary metastasis with complex fistula. Its minimally invasive and repeatability can help to reduce the frequency of repeated hospitalization and the risk of infection, save medical resources, and provide new ideas for the exploration of multimodal embolization techniques in interventional medicine, which has a profound impact on improving the quality of life of patients with end-stage cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient was diagnosed with osteosarcoma by histology or cytology, and pulmonary metastasis with bronchopleural fistula (BPF) was confirmed by imaging (CT/PET-CT);
* Present with clinical symptoms associated with BPF (e.g., hemoptysis, pneumothorax, persistent pleural infection, etc.) that are ineffective or poorly responded to traditional treatments (pharmacologic hemostasis, closed thoracic drainage);
* Angiographically confirmed abnormal bronchial or intercostal artery blood supply to the fistula and anatomy suitable for NBCA with coil embolization;
* Age ≤75 years, ECOG performance status ≤2, and predicted survival ≥3 months.
* Coagulation function was basically normal.

Exclusion Criteria:

* Had a history of severe allergy or contraindication to NBCA glue, iodine contrast agent or coil materials;
* Severe cardiopulmonary dysfunction (e.g., NYHA class III-IV, FEV1 < 30% predicted, uncontrolled pulmonary hypertension);
* Angiographic abnormalities of the target vessel anatomy (e.g., severe tortuosity, stenosis, or occlusion) prevented the catheter from safely reaching the target embolization site;
* Active systemic infection (e.g., sepsis, active tuberculosis) or uncontrolled local infection;
* Other major organ failure (Child-Pugh C cirrhosis, eGFR < 30 mL/min/1.73m²);
* Women who are pregnant or lactating or plan to become pregnant during the study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 1, 2019 to December 31, 2023, patients with pulmonary metastasis of osteosarcoma complicated with BPLF who underwent interventional treatment in the hospital were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
OS，Overall Survival | From the time of treatment to the death from any cause, assessed up to 50 months.
  The patient received treatment until death.
PFS，Progress Free Survival | From the time of treatment to tumor progression or date of death from any cause, whichever came first, assessed up to 50 months
  Time of progression or death of the patient.

IPD SHARING:
Plan to Share IPD: No